CLINICAL TRIAL: NCT02791516
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Study to Compare the Efficacy and Safety of Romosozumab With Placebo in Postmenopausal South Korean Women With Osteoporosis
Brief Title: A Safety and Efficacy Study to Evaluate Romosozumab (AMG 785) in South Korean Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20150242
Record Dates: First submitted 2016-06-02; First posted 2016-06-06 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis.; Osteoporosis-Postmenopausal.; Bone Diseases-Metabolic.; Bone Diseases.; Musculoskeletal Diseases.
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic; Bone Diseases; Musculoskeletal Diseases | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once a month for 6 months.
  Interventions: Drug: Placebo
- Romosozumab (Experimental): Participants received 210 mg romosozumab by subcutaneous injection once a month for 6 months.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection once a month (QM)
  Other Names: AMG 785; Evenity
  Arms: Romosozumab
Drug: Placebo — Administered by subcutaneous injections once a month
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the effect of treatment with romosozumab for 6 months compared with placebo on percent changes in bone mineral density (BMD) at the lumbar spine as assessed by dual-energy X-ray absorptiometry (DXA) in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal Korean women, ≥ 55 to ≤ 90 years of age at enrollment.
* Postmenopause is defined as no spontaneous vaginal bleeding or spotting for 12 or more consecutive months prior to screening.
* BMD T-score </= -2.50 at the lumbar spine, total hip or femoral neck.
* At least 2 vertebrae in the L1 through L4 region and at least one hip are evaluable by DXA.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Subjects with a BMD T-score </= -4.0 at the lumbar spine, total hip, or femoral neck.
* History of hip fracture.
* Bone disease other than osteoporosis/ or evidence of any other clinically significant disorder, condition/ or disease or significant laboratory abnormalities.
* Known sensitivity or intolerance calcium and vitamin D products.
* Other exclusion criteria may apply.

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- South Korea (6):
  - Research Site, Busan
  - Research Site, Gwangju
  - Research Site, Namdong-gu, Incheon
  - Research Site, Seongnam Si Gyeonggi Do
  - Research Site, Seoul
  - Research Site, Suwon-si, Gyeonggi-do

REFERENCES:
- [Derived] Baek KH, Chung YS, Koh JM, Kim IJ, Kim KM, Min YK, Park KD, Dinavahi R, Maddox J, Yang W, Kim S, Lee SJ, Cho H, Lim SK. Romosozumab in Postmenopausal Korean Women with Osteoporosis: A Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study. Endocrinol Metab (Seoul). 2021 Feb;36(1):60-69. doi: 10.3803/EnM.2020.848. Epub 2021 Feb 24. PMID 33677928
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 centers in South Korea. Participants were enrolled from 16 January 2017 to 17 August 2017.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either romosozumab 210 mg subcutaneously (SC) QM or matched placebo SC QM. Upon completion of the 6-month treatment period, participants were followed for an additional 3 months.
Groups:
- Romosozumab 210 mg: Participants received 210 mg romosozumab by subcutaneous injection once a month for 6 months.
Period: Overall Study
Arm/Group | Placebo | Romosozumab 210 mg
Started | 33 | 34
Completed 6-month Treatment Period | 33 | 33
Completed (Completed 9-month study period) | 32 | 33
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 210 mg | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.2) | 66.7 (7.6) | 67.5 (7.4)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 13 | 14 | 27
  ≥ 65 to < 75 years | 13 | 16 | 29
  ≥ 75 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 33 | 34 | 67
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: T-score] — The T-score is a comparison of a person's bone density with that of a healthy 30-year-old of the same sex. Lower scores (more negative) mean lower bone density: A T-score of -2.5 or lower qualifies as osteoporosis and a T-score of -1.0 to - 2.5 signifies osteopenia, meaning below-normal bone density without full osteoporosis.
  T-score | -2.6483 (0.6450) | -2.6622 (0.8155) | -2.6554 (0.7310)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] — The T-score is a comparison of a person's bone density with that of a healthy 30-year-old of the same sex. Lower scores (more negative) mean lower bone density: A T-score of -2.5 or lower qualifies as osteoporosis and a T-score of -1.0 to - 2.5 signifies osteopenia, meaning below-normal bone density without full osteoporosis.
  T-score | -2.1797 (0.6243) | -2.1515 (0.7114) | -2.1654 (0.6650)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] — The T-score is a comparison of a person's bone density with that of a healthy 30-year-old of the same sex. Lower scores (more negative) mean lower bone density: A T-score of -2.5 or lower qualifies as osteoporosis and a T-score of -1.0 to - 2.5 signifies osteopenia, meaning below-normal bone density without full osteoporosis
  T-score | -2.5309 (0.5395) | -2.4494 (0.6069) | -2.4896 (0.5718)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 6 in Bone Mineral Density at the Lumbar Spine
Description: Bone mineral density (BMD) at the lumbar spine was assessed by dual-energy x-ray absorptiometry (DXA). Images were assessed by a central reader.
Time Frame: Baseline and month 6
Population: Randomized participants who had a baseline DXA BMD measurement and at least 1 postbaseline DXA BMD measurement at the lumbar spine.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 31 | 33
percent change | -0.1 (0.8) | 9.5 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model adjusting for treatment, baseline DXA BMD value, machine type, and machine type-by-baseline DXA BMD value; LS Mean Difference = 9.6, 95% CI 2-sided [7.6 to 11.5], Standard Error of Mean 1.0

2. Secondary Outcome: Percent Change From Baseline to Month 6 in Bone Mineral Density at the Total Hip
Description: Bone mineral density (BMD) at the total hip was assessed by dual-energy x-ray absorptiometry (DXA). Images were assessed by a central reader.
Time Frame: Baseline and month 6
Population: Randomized participants who had a baseline DXA BMD measurement and at least 1 postbaseline DXA BMD measurement at the total hip.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 31 | 33
percent change | 0.3 (0.4) | 2.9 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model adjusting for treatment, baseline DXA BMD value, machine type, and machine type-by-baseline DXA BMD value; LS Mean Difference = 2.6, 95% CI 2-sided [1.4 to 3.7], Standard Error of Mean 0.6

3. Secondary Outcome: Percent Change From Baseline to Month 6 in Bone Mineral Density at the Femoral Neck
Description: Bone mineral density (BMD) at the femoral neck was assessed by dual-energy x-ray absorptiometry (DXA). Images were assessed by a central reader.
Time Frame: Baseline and month 6
Population: Randomized participants who had a baseline DXA BMD measurement and at least 1 postbaseline DXA BMD measurement at the femoral neck.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 31 | 33
percent change | 0.8 (0.7) | 3.0 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority; p = 0.004, ANCOVA; ANCOVA model adjusting for treatment, baseline DXA BMD value, machine type, and machine type-by-baseline DXA BMD value; LS Mean Difference = 2.2, 95% CI 2-sided [0.7 to 3.6], Standard Error of Mean 0.7

ADVERSE EVENTS:
Time Frame: 9 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romosozumab 210 mg
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/34
Other Adverse Events (participants affected / at risk) | 4/33 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Romosozumab 210 mg (N=34)
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Romosozumab 210 mg (N=34)
Nasopharyngitis (Infections and infestations) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT02791516/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT02791516/SAP_001.pdf